CLINICAL TRIAL: NCT06036667
Title: Safety and Efficacy of Coaxial Smart Drain (Redax TM) in Uniportal-VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID 2388
Record Dates: First submitted 2023-02-21; First posted 2023-09-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pleural Effusion; Video Assisted Thoracic Surgery; Chest Tubes
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group (Experimental): All patients undergone Uniportal-VATS upper lobectomy with 28Fr Smart Coaxial drain placed at the end of surgery
  Interventions: Procedure: 28Fr "coaxial smart drain" chest tube
- Study group 1 (No Intervention): All patients undergone Uniportal-VATS upper lobectomy with standard 28Fr chest drain placed at the end of surgery
- Study group 2 (Experimental): All patients undergone Biportal-VATS upper lobectomy with 28Fr Smart Coaxial drain placed at the end of surgery
  Interventions: Procedure: 28Fr "coaxial smart drain" chest tube

INTERVENTIONS:
Procedure: 28Fr "coaxial smart drain" chest tube — To evaluate the efficacy of one 28Fr chest tube ("coaxial smart drain" versus standard chest tube according to local practice, types of drainage availability in each centre, surgeon's choice etc) after Uniportal- or Biportal-VATS upper lobectomies.
  Arms: Study group; Study group 2

SUMMARY:
The aim of the study is to evaluate efficacy and safety of "Smart Coaxial drain" (Redax TM, Poggio Rusco, Mantova, Italia) in terms of total amount of effusion drained, incidence of residual effusion at Chest X-Ray and patient's comfort in Uniportal- and Biportal-VATS upper lobectomies.

In particular, to evaluate in Uniportal-VATS upper lobectomies the efficacy and safety of smart coaxial drains compared with standard silicone chest tubes.

DETAILED DESCRIPTION:
At the end of lung surgery, usually surgeons placed one or more chest tubes. There are several types of chest tubes and the type used by surgeons depends on centre avaiability/ local practice or surgeon choice etc...Coaxial smart drains are used in clinical practice since several years in Thoracic Surgery. In thoracoscopic (VATS) surgery usually only one chest tube is placed. In this study, we evaluate the efficacy of placement of 28Fr "coaxial smart drain" chest tube versus 28 Fr standard chest tube after Uniportal- or Biportal-VATS upper lobectomies in terms of total amount of effusion drained, incidence of residual effusion at Chest X-Ray and patient's confort.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone upper right or left lobectomy in Uniportal- or Biportal-VATS

Exclusion Criteria:

* Patients undergone open surgery
* Patients undergone middle or lower lobectomies
* Patients undergone chest wall/or wedge resections

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Fluid output 1 | At 24 hours from surgery
  Total fluid amount
Fluid output 2 | At 48 hours from surgery
  Total fluid amount
Fluid output 3 | At 72 hours from surgery
  Total fluid amount
Fluid output 4 | At 96 hours from surgery
  Total fluid amount
Residual pleural effusion at chest X-Ray | 72 hours after surgery
  Residual pleural effusion at chest X-Ray before chest tube removal. The entity of pleural effusion is measured as "intercostal spaces", counted on posterior costal arches
subcutaneous emphysema 1 | At 24 hours after surgery
  incidence of subcutaneous emphysema
subcutaneous emphysema 2 | At 48 hours after surgery
  incidence of subcutaneous emphysema
subcutaneous emphysema 3 | At 72 hours after surgery
  incidence of subcutaneous emphysema

SECONDARY OUTCOMES:
Tube obstruction | during chest tube removal procedure
  tube obstructed by blood clots
Pain related to chest tube 1 | At 24 hours after surgery
  Pain measured in each postoperative day on VAS scale (Visual Analogue Scale, range:from 0 to 10; VAS>4 and <10 indicates moderate to severe pain)
Pain related to chest tube 2 | At 48 hours after surgery
  Pain measured in each postoperative day on VAS scale (Visual Analogue Scale, range:from 0 to 10; VAS>4 and <10 indicates moderate to severe pain)
Pain related to chest tube 3 | At 72 hours after surgery
  Pain measured in each postoperative day on VAS scale (Visual Analogue Scale, range:from 0 to 10; VAS>4 and <10 indicates moderate to severe pain)
Pain related to chest tube 4 | At 96 hours after surgery
  Pain measured in each postoperative day on VAS scale (Visual Analogue Scale, range:from 0 to 10; VAS>4 and <10 indicates moderate to severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Dania Nachira, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No